CLINICAL TRIAL: NCT05131971
Title: A Randomized, Double-Blind, Placebo Controlled, Single Dose Escalation Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of GSK3888130B in Healthy Participants Aged 18-55 Inclusive
Brief Title: A Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics (PD) of GSK3888130B in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 213960; 2021-002063-22 (EudraCT Number)
Record Dates: First submitted 2021-10-27; First posted 2021-11-23 (Actual); Results first posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis; Colitis, Ulcerative
Keywords: Anti-Drug Antibodies; Double-blind; GSK3888130B; Pharmacodynamics; Pharmacokinetics; Single Dose Escalation
MeSH Terms: conditions — Multiple Sclerosis; Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive either GSK3888130B or placebo in single ascending dose cohorts.
Who Masked: Participant, Investigator
Masking Description: This will be a double-blind study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- Cohort 1: Participants receiving GSK3888130B at dose level 1 (Experimental)
  Interventions: Drug: GSK3888130B
- Cohort 1: Participants receiving placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Cohort 2: Participants receiving GSK3888130B at dose level 2 (Experimental)
  Interventions: Drug: GSK3888130B
- Cohort 2: Participants receiving placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Cohort 3: Participants receiving GSK3888130B at dose level 3 (Experimental)
  Interventions: Drug: GSK3888130B
- Cohort 3: Participants receiving placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Cohort 4: Participants receiving GSK3888130B at dose level 4 (Experimental)
  Interventions: Drug: GSK3888130B
- Cohort 4: Participants receiving placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Cohort 5: Participants receiving GSK3888130B at dose level 5 (Experimental)
  Interventions: Drug: GSK3888130B
- Cohort 5: Participants receiving placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Cohort 6: Participants receiving GSK3888130B at dose level 6 (Experimental)
  Interventions: Drug: GSK3888130B
- Cohort 6: Participants receiving placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Cohort 7: Participants receiving GSK3888130B at dose level 7 (Experimental)
  Interventions: Drug: GSK3888130B
- Cohort 7: Participants receiving placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK3888130B — GSK3888130B will be administered.
  Arms: Cohort 1: Participants receiving GSK3888130B at dose level 1; Cohort 2: Participants receiving GSK3888130B at dose level 2; Cohort 3: Participants receiving GSK3888130B at dose level 3; Cohort 4: Participants receiving GSK3888130B at dose level 4; Cohort 5: Participants receiving GSK3888130B at dose level 5; Cohort 6: Participants receiving GSK3888130B at dose level 6; Cohort 7: Participants receiving GSK3888130B at dose level 7
Drug: Placebo — Placebo will be administered.
  Arms: Cohort 1: Participants receiving placebo; Cohort 2: Participants receiving placebo; Cohort 3: Participants receiving placebo; Cohort 4: Participants receiving placebo; Cohort 5: Participants receiving placebo; Cohort 6: Participants receiving placebo; Cohort 7: Participants receiving placebo

SUMMARY:
This is a first time in human study designed to assess the safety, tolerability, pharmacokinetics and PD of GSK3888130B over a range of dose levels in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 55 years of age inclusive.
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* Participants with a confirmed positive vaccination status for Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) vaccines administered at least 30 days prior to dosing in the study.
* SARS-CoV-2 screening test negative as per local guidance.
* Participants with history of current/seasonal vaccination status for influenza or who consent to receive influenza vaccine at least 30 days prior to dosing, if study dosing is during influenza season (1st October to 30th April).
* Body weight greater than or equal to (>=) 50 kilograms (kg) and body mass index (BMI) within the range 19.5-32 kilograms per square meter (kg/m^2) (inclusive).
* Male and/or female of non-childbearing potential
* Capable of giving signed informed consent.

Exclusion Criteria:

* Prior medical history of anaphylaxis.
* Immunodeficiency or autoimmunity assessed by medical history.
* A history of recurrent infections.
* Treatment of a chronic infection within 3 months prior to the first dose of study drug.
* Any acute infection (including upper respiratory tract infections and urinary tract infections) which has not fully resolved within four weeks of dosing
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy.
* Current or chronic history of liver disease or known hepatic or biliary abnormalities.
* Participants with a history of renal disease or renal abnormalities.
* A clinically significant abnormality in the 12-lead ECG performed at screening.
* A clinically significant abnormality in the Holter monitor performed at screening.
* History of malignancy, including malignant or non-malignant skin cancer.
* Participants with known SARS-CoV-2 positive contacts in the past 14 days.
* Prior moderate/severe SARS-CoV-2 infection requiring oxygen supplementation or admission to hospital.
* Antibiotics or antiviral therapy within 30 days of dosing.
* Receipt of live vaccination within 30 days of dosing or plan to receive live vaccination during the study.
* Use of prescription drugs or non-prescription drugs, including non-steroidal anti inflammatory drug (NSAIDs), within 7 days prior to dosing, if in the opinion of the Investigator (in consultation with the GlaxoSmithKline [GSK] Medical Monitor if required) the medication will interfere with the study procedures or compromise participant safety.
* The participant has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day of the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than 4 new chemical entities within 12 months prior to dosing.
* A positive drug/alcohol test at screening or Day -1
* The participant is at high-risk of Mycobacterium tuberculosis (MTB) infection in the opinion of the Investigator.
* History of asthma, allergic rhinitis or atopic dermatitis defined by the need for intermittent or continuous therapy or any other significant allergies that, in the opinion of the investigator contraindicates their participation.
* History of severe adverse reaction to local anesthetic.
* Presence of keloids or history of keloids.
* Prothrombin time (PT) or activated partial thromboplastin time (aPTT) >1.5x upper limit of normal (ULN) at screening.
* History or presence of excessive bleeding or coagulation disorders that in the opinion of the Investigator poses a safety risk with regards to participation in the trial.
* Presence of tattoos, naevi or other skin abnormalities on the volar forearm Fitzpatrick skin color grades V in the opinion of the investigator, interfere with study assessments
* Participating, within 7 days of dosing, in recreational sun-bathing, or use of sunbed, on the area of the skin from wrist to shoulder inclusive.
* Current smoker or user of tobacco- or nicotine-containing products (e.g. nicotine patches or vaporizing devices) during or within 30 days prior to study participation.
* An average weekly intake of >14 units of alcohol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-10-12 (Actual); Study Completion 2023-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total 54 participants were enrolled in this study. Placebo arms were combined as pre-specified in reporting and analysis plan. Dosing information (dosage strengths) has not been disclosed as it is considered as company confidential information (CCI). Dose levels are presented as Dose levels 1 to 7 along with directionality of the dosage within each arm/group.
Groups:
- Placebo: Participants received a placebo matching GSK3888130B either intravenous (IV) infusion or subcutaneous (SC) injection on Day 1.
- GSK3888130B Dose Level 1 IV: Participants received a single dose of GSK3888130B dose level 1, intravenous (IV) infusion on Day 1. Dose level 1 is the lowest dose level.
- GSK3888130B Dose Level 2 IV: Participants received a single dose of GSK3888130B dose level 2, IV infusion on Day 1. Dose level 2 is greater than dose level 1.
- GSK3888130B Dose Level 3 SC: Participants received a single dose of GSK3888130B dose level 3, subcutaneous (SC) injection on Day 1. Dose level 3 is greater than dose level 2.
- GSK3888130B Dose Level 4 IV: Participants received a single dose of GSK3888130B dose level 4, IV infusion on Day 1. Dose level 4 is greater than dose level 3.
- GSK3888130B Dose Level 5 SC: Participants received a single dose of GSK3888130B dose level 5, SC injection on Day 1. Dose level 5 is greater than dose level 4.
- GSK3888130B Dose Level 6 IV: Participants received a single dose of GSK3888130B dose level 6, IV infusion on Day 1. Dose level 6 is greater than dose level 5.
- GSK3888130B Dose Level 7 IV: Participants received a single dose of GSK3888130B dose level 7, IV infusion on Day 1. Dose level 7 is the highest dose level.
Period: Overall Study
Arm/Group | Placebo | GSK3888130B Dose Level 1 IV | GSK3888130B Dose Level 2 IV | GSK3888130B Dose Level 3 SC | GSK3888130B Dose Level 4 IV | GSK3888130B Dose Level 5 SC | GSK3888130B Dose Level 6 IV | GSK3888130B Dose Level 7 IV
Started | 15 | 3 | 3 | 6 | 6 | 6 | 9 | 6
Completed | 15 | 3 | 3 | 6 | 6 | 6 | 9 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Placebo arms were combined as pre-specified in reporting and analysis plan.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK3888130B Dose Level 1 IV | GSK3888130B Dose Level 2 IV | GSK3888130B Dose Level 3 SC | GSK3888130B Dose Level 4 IV | GSK3888130B Dose Level 5 SC | GSK3888130B Dose Level 6 IV | GSK3888130B Dose Level 7 IV | Total
Number analyzed (Participants) | 15 | 3 | 3 | 6 | 6 | 6 | 9 | 6 | 54
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 40.3 (8.93) | 40.0 (7.94) | 48.3 (3.06) | 38.8 (8.75) | 41.2 (9.52) | 40.8 (7.70) | 38.7 (9.86) | 41.5 (11.57) | 40.6 (8.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 15 | 3 | 3 | 6 | 6 | 6 | 9 | 6 | 54
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — The "All Other Races" category (ASIAN, WHITE and MIXED RACE where 0<n<11) are combined into one category to maintain participant confidentiality and privacy.
  Participants
    All Other Races | 15 | 3 | 3 | 6 | 6 | 6 | 9 | 6 | 54

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is any serious adverse event that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or any other situation according to medical or scientific judgment.
Time Frame: Up to 160 days
Population: Safety Population included all participants who received study intervention. Placebo arms were combined as pre-specified in reporting and analysis plan.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3888130B Dose Level 1 IV | GSK3888130B Dose Level 2 IV | GSK3888130B Dose Level 3 SC | GSK3888130B Dose Level 4 IV | GSK3888130B Dose Level 5 SC | GSK3888130B Dose Level 6 IV | GSK3888130B Dose Level 7 IV
Number analyzed (Participants) | 15 | 3 | 3 | 6 | 6 | 6 | 9 | 6
Participants
  AEs | 8 | 3 | 2 | 6 | 2 | 4 | 8 | 5
  SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Clinically Significant Changes in Hematology Results
Description: Blood samples were collected for analysis of following hematology parameters: Basophils, Eosinophils, Hematocrit, Hemoglobin (Hg), Lymphocytes, Mean corpuscular Hg, Mean corpuscular volume, Monocytes, Platelet count, Red blood cell count, Reticulocytes, Total Neutrophils, and White blood cells count (WBC). Number of participants with clinically significant changes in hematology were reported. Clinical significance was determined by the investigator.
Time Frame: Up to 85 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3888130B Dose Level 1 IV | GSK3888130B Dose Level 2 IV | GSK3888130B Dose Level 3 SC | GSK3888130B Dose Level 4 IV | GSK3888130B Dose Level 5 SC | GSK3888130B Dose Level 6 IV | GSK3888130B Dose Level 7 IV
Number analyzed (Participants) | 15 | 3 | 3 | 6 | 6 | 6 | 9 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Worst-case Cluster of Differentiation (CD) 4+ T Cell Counts Results by Maximum Grade Increase Post-Baseline Relative to Baseline
Description: Blood samples were collected for the analysis of CD4+ T Cell Counts. The CD4+ T Cell Counts were graded according to National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE). Grade 0: Above 0.5*10^9 cells/Liter (L), Grade 1: <0.5 to 0.2*10^9 cells/L, Grade 2: <0.2 to 0.05*10^9 cells/L, Grade 3: Below 0.05*10^9 cells/L. Baseline was defined as the latest pre-dose assessment. An increase was defined as an increase in grade relative to Baseline grade. Any worst-case post Baseline increase to Grade 1, Grade 2 and Grade 3 are presented.
Time Frame: Baseline (Day 1) and up to 85 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3888130B Dose Level 1 IV | GSK3888130B Dose Level 2 IV | GSK3888130B Dose Level 3 SC | GSK3888130B Dose Level 4 IV | GSK3888130B Dose Level 5 SC | GSK3888130B Dose Level 6 IV | GSK3888130B Dose Level 7 IV
Number analyzed (Participants) | 15 | 3 | 3 | 6 | 6 | 6 | 9 | 6
Participants
  Increase to Grade 1 | 4 | 1 | 1 | 1 | 1 | 3 | 5 | 4
  Increase to Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Worst-case Creatinine Results by Maximum Grade Increase Post-Baseline Relative to Baseline
Description: Blood samples were collected for the analysis of Creatinine. Creatinine was graded according to the NCI-CTCAE. Grade 0: <1.5* Baseline, or increase from Baseline <26 micromoles per liter (umol/L), Grade 1: 1.5 to 1.9* Baseline, or increase from Baseline >=26 umol/L, Grade 2: 2.0 to 2.9* Baseline, Grade 3: >=3.0* Baseline, or >=354 umol/L. Baseline was defined as the latest pre-dose assessment. An increase was defined as an increase in grade relative to Baseline grade. Any worst-case post Baseline increase to Grade 1, Grade 2 and Grade 3 are presented.
Time Frame: Baseline (Day 1) and up to 85 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3888130B Dose Level 1 IV | GSK3888130B Dose Level 2 IV | GSK3888130B Dose Level 3 SC | GSK3888130B Dose Level 4 IV | GSK3888130B Dose Level 5 SC | GSK3888130B Dose Level 6 IV | GSK3888130B Dose Level 7 IV
Number analyzed (Participants) | 15 | 3 | 3 | 6 | 6 | 6 | 9 | 6
Participants
  Increase to Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Increase to Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Clinically Significant Changes in Clinical Chemistry Results
Description: Blood samples were collected for analysis of following clinical chemistry parameters: Alanine Aminotransferase, Alkaline Phosphatase, Aspartate Aminotransferase, Calcium, Total and Direct bilirubin, Glucose, Potassium, Sodium, Total protein, Lactate dehydrogenase, Haptoglobins and Urea. Number of participants with clinically significant changes in clinical chemistry were reported. Clinical significance was determined by the investigator.
Time Frame: Up to 85 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3888130B Dose Level 1 IV | GSK3888130B Dose Level 2 IV | GSK3888130B Dose Level 3 SC | GSK3888130B Dose Level 4 IV | GSK3888130B Dose Level 5 SC | GSK3888130B Dose Level 6 IV | GSK3888130B Dose Level 7 IV
Number analyzed (Participants) | 15 | 3 | 3 | 6 | 6 | 6 | 9 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Worst-case Any Increase in Urinalysis Results Post-Baseline Relative to Baseline
Description: Urine samples were collected for analysis of Specific gravity, potential of hydrogen (pH), glucose, protein, erythrocytes, ketones, bilirubin, urobilinogen, nitrite, and leukocyte in urine by dipstick. The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameters can be read as negative, trace, 1+, 2+, 3+ indicating proportional concentrations in the urine sample. Any increase means any increase to trace, 1+, 2+ or 3+ post-Baseline relative to Baseline. Baseline was defined as the latest pre-dose assessment. Number of participants with worst-case any increase in urinalysis results post-Baseline relative to Baseline has been presented.
Time Frame: Baseline (Day 1) and up to 85 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3888130B Dose Level 1 IV | GSK3888130B Dose Level 2 IV | GSK3888130B Dose Level 3 SC | GSK3888130B Dose Level 4 IV | GSK3888130B Dose Level 5 SC | GSK3888130B Dose Level 6 IV | GSK3888130B Dose Level 7 IV
Number analyzed (Participants) | 15 | 3 | 3 | 6 | 6 | 6 | 9 | 6
Participants
  Bilirubin | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Erythrocytes | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0
  Glucose | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Ketones | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Leukocytes | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nitrite | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Protein | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Specific Gravity | 8 | 3 | 2 | 4 | 5 | 6 | 5 | 6
  Urobilinogen | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  pH | 12 | 3 | 2 | 5 | 4 | 6 | 8 | 5

7. Primary Outcome: Number of Participants With Clinically Significant Changes in Vital Sign Results
Description: Vital signs included systolic and diastolic blood pressure, pulse and respiratory rate and were measured with the participant in semi-supine position after 5 minutes rest. Temperature was also measured as a vital sign but did not require positioning or rest prior to measuring. Clinical significance was determined by the investigator.
Time Frame: Up to 85 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3888130B Dose Level 1 IV | GSK3888130B Dose Level 2 IV | GSK3888130B Dose Level 3 SC | GSK3888130B Dose Level 4 IV | GSK3888130B Dose Level 5 SC | GSK3888130B Dose Level 6 IV | GSK3888130B Dose Level 7 IV
Number analyzed (Participants) | 15 | 3 | 3 | 6 | 6 | 6 | 9 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With Positive Cytomegalovirus (CMV) Deoxyribonucleic Acid (DNA) and Varicella Zoster Virus (VZV) DNA
Description: VZV-Nucleic acid from blood samples were extracted using the QIASymphony SP followed by TaqMan real time polymerase chain reaction (PCR) for amplification and detection. Murine cytomegalovirus (mCMV) was used as an internal control (IC) and was introduced during the extraction process. CMV-Nucleic acid was extracted using the QIASymphony SP/AS followed by automated set up of Artus real time PCR using the Rotor-Gene Q for amplification and detection. Baseline was defined as the latest pre-dose assessment. Number of participants with Positive CMV DNA and VZV DNA has been presented.
Time Frame: Baseline (Day 1), Day 15 and Day 85
Population: Safety Population included all participants who received study intervention. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the 'Overall Number of Participants Analyzed' field. 'Number Analyzed' signifies participants evaluable for the specified time points. Placebo arms were combined as pre-specified in reporting and analysis plan.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3888130B Dose Level 1 IV | GSK3888130B Dose Level 2 IV | GSK3888130B Dose Level 3 SC | GSK3888130B Dose Level 4 IV | GSK3888130B Dose Level 5 SC | GSK3888130B Dose Level 6 IV | GSK3888130B Dose Level 7 IV
Number analyzed (Participants) | 15 | 3 | 3 | 6 | 6 | 6 | 9 | 6
Participants
  Cytomegalovirus DNA, Baseline (Day 1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cytomegalovirus DNA, Day 15: number analyzed (Participants) | 15 | 2 | 3 | 6 | 6 | 6 | 9 | 6
  Cytomegalovirus DNA, Day 15 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cytomegalovirus DNA, Day 85 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Varicella Zoster Virus DNA, Baseline (Day 1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Varicella Zoster Virus DNA, Day 15: number analyzed (Participants) | 15 | 2 | 3 | 6 | 6 | 6 | 9 | 6
  Varicella Zoster Virus DNA, Day 15 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Varicella Zoster Virus DNA, Day 85 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Participants With Positive Epstein-Barr Virus (EBV) DNA
Description: EBV DNA was assessed and qualitative data has been presented. Data has been categorized into 'Positive >=LLQ' and 'Positive < LLQ'. LLQ is lower limit of quantification. Participants who had EBV DNA values >=LLQ were categorized as 'Positive >=LLQ'. This represents a positive result that is above the assay limit of quantification. Participants who had EBV DNA values <LLQ were categorized as 'Positive <LLQ'. This represents a positive result that is below the assay limit of quantification. Baseline was defined as the latest pre-dose assessment.
Time Frame: Baseline (Day 1), Day 15 and Day 85
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3888130B Dose Level 1 IV | GSK3888130B Dose Level 2 IV | GSK3888130B Dose Level 3 SC | GSK3888130B Dose Level 4 IV | GSK3888130B Dose Level 5 SC | GSK3888130B Dose Level 6 IV | GSK3888130B Dose Level 7 IV
Number analyzed (Participants) | 15 | 3 | 3 | 6 | 6 | 6 | 9 | 6
Participants
  Baseline (Day 1), Positive < LLQ | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
  Baseline (Day 1), Positive >= LLQ | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Day 15, Positive < LLQ: number analyzed (Participants) | 15 | 2 | 3 | 6 | 6 | 6 | 9 | 6
  Day 15, Positive < LLQ | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
  Day 15, Positive >= LLQ: number analyzed (Participants) | 15 | 2 | 3 | 6 | 6 | 6 | 9 | 6
  Day 15, Positive >= LLQ | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Day 85, Positive < LLQ | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 85, Positive >= LLQ | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1

10. Primary Outcome: Number of Participants With Worst-case Post-Baseline Abnormal Electrocardiogram (ECG) Findings
Description: Twelve lead ECGs were obtained using an ECG machine that automatically calculated the heart rate and measured PR, QRS, QT, and QT corrected interval. Abnormal findings were categorized as clinically significant (CS) and not clinically significant (NCS). Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Data for number of participants with worst case post-Baseline abnormal ECG findings have been presented.
Time Frame: Up to 85 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3888130B Dose Level 1 IV | GSK3888130B Dose Level 2 IV | GSK3888130B Dose Level 3 SC | GSK3888130B Dose Level 4 IV | GSK3888130B Dose Level 5 SC | GSK3888130B Dose Level 6 IV | GSK3888130B Dose Level 7 IV
Number analyzed (Participants) | 15 | 3 | 3 | 6 | 6 | 6 | 9 | 6
Participants
  CLINICALLY SIGNIFICANT | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  NOT CLINICALLY SIGNIFICANT | 12 | 1 | 2 | 6 | 4 | 6 | 7 | 5

11. Secondary Outcome: Serum Concentrations of GSK3888130B for Dose Levels 1, 2 and 4 Intravenous Administration
Description: Blood samples were collected at indicated time points for measurement of serum concentrations of GSK3888130B following intravenous administration. Pharmacokinetic (PK) Population consisted of all participants in the Safety analysis set who had received an active study intervention and had at least 1 non-missing post dose PK assessment (Non-quantifiable [NQ] values were considered as non-missing values).
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 4, 8, 12, 24, 48 hours; Days 6, 8, 10, 15, 21, 29, 57, and 85
Population: PK Population. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the 'Overall Number of Participants Analyzed' field. 'Number Analyzed' signifies participants evaluable for the specified time points.
Measure: Geometric Mean (95% Confidence Interval); unit: Nanograms per milliliter (ng/mL)
Arm/Group | GSK3888130B Dose Level 1 IV | GSK3888130B Dose Level 2 IV | GSK3888130B Dose Level 4 IV
Number analyzed (Participants) | 3 | 3 | 6
Nanograms per milliliter (ng/mL)
  DAY 1 (Pre-dose) | NA [NA to NA] — Geometric mean and 95% CI could not be calculated if any values were imputed due to being non-quantifiable (NQ). | NA [NA to NA] — Geometric mean and 95% CI could not be calculated if any values were imputed due to being NQ. | NA [NA to NA] — Geometric mean and 95% CI could not be calculated if any values were imputed due to being NQ.
  DAY 1 (15 Minutes) | 363.2 [196.7 to 670.9] | 2155.9 [1003.0 to 4634.4] | 15901.1 [13993.4 to 18069.0]
  DAY 1 (30 Minutes) | 893.1 [504.7 to 1580.5] | 4717.5 [3173.3 to 7013.1] | 35633.0 [30628.5 to 41455.2]
  DAY 1 (4 Hours) | 761.4 [677.2 to 856.1] | 4497.0 [2542.8 to 7953.0] | 32762.8 [28319.4 to 37903.3]
  DAY 1 (8 Hours) | 753.5 [483.7 to 1173.8] | 3964.2 [1974.7 to 7958.0] | 31180.8 [27855.3 to 34903.4]
  DAY 1 (12 Hours) | 758.1 [601.3 to 955.8] | 3599.9 [2601.7 to 4981.2] | 29821.8 [26986.2 to 32955.3]
  DAY 1 (24 Hours) | 720.8 [558.6 to 930.0] | 3781.5 [2095.7 to 6823.7] | 28096.6 [26173.0 to 30161.6]
  DAY 1 (48 Hours) | 572.8 [401.3 to 817.7] | 3184.0 [2280.6 to 4445.1] | 23358.3 [20418.2 to 26721.8]
  DAY 6 | NA [NA to NA] — Geometric mean and 95% CI could not be calculated if any values were imputed due to being NQ. | 2134.0 [1229.6 to 3703.5] | 15978.7 [14176.6 to 18009.9]
  DAY 8 | NA [NA to NA] — Geometric mean and 95% CI could not be calculated if any values were imputed due to being NQ. | 1862.5 [883.6 to 3926.1] | 14071.9 [13088.2 to 15129.5]
  DAY 10: number analyzed (Participants) | 2 | 3 | 6
  DAY 10 | NA [NA to NA] — Geometric mean and 95% CI could not be calculated if any values were imputed due to being NQ. | 1850.1 [928.4 to 3687.1] | 12873.0 [11718.1 to 14141.7]
  DAY 15: number analyzed (Participants) | 2 | 3 | 6
  DAY 15 | NA [NA to NA] — Geometric mean and 95% CI could not be calculated if any values were imputed due to being NQ. | 1539.6 [740.1 to 3202.8] | 10293.7 [9018.8 to 11748.8]
  DAY 21: number analyzed (Participants) | 3 | 3 | 5
  DAY 21 | NA [NA to NA] — Geometric mean and 95% CI could not be calculated if any values were imputed due to being NQ. | 1263.0 [416.5 to 3829.5] | 8485.9 [7647.8 to 9415.9]
  DAY 29 | NA [NA to NA] — Geometric mean and 95% CI could not be calculated if any values were imputed due to being NQ. | 1027.3 [404.7 to 2607.4] | 6904.9 [5741.6 to 8304.0]
  DAY 57 | NA [NA to NA] — Geometric mean and 95% CI could not be calculated if any values were imputed due to being NQ. | 625.4 [192.9 to 2027.2] | 3545.2 [2721.4 to 4618.4]
  DAY 85 | NA [NA to NA] — Geometric mean and 95% CI could not be calculated if any values were imputed due to being NQ. | NA [NA to NA] — Geometric mean and 95% CI could not be calculated if any values were imputed due to being NQ. | 1797.5 [1152.8 to 2802.8]

12. Secondary Outcome: Serum Concentrations of GSK3888130B for Dose Levels 3 and 5 Subcutaneous Administration
Description: Blood samples were collected at indicated time points for measurement of serum concentrations of GSK3888130B following subcutaneous administration.
Time Frame: Day 1: Pre-dose, 4, 8, 12, 24, 48 hours; Days 6, 8, 10, 15, 21, 29, 57, and 85
Population: Pharmacokinetic Population consisted of all participants in the Safety analysis set who had received an active study intervention and had at least 1 non-missing post dose PK assessment (Non-quantifiable [NQ] values were considered as non-missing values).
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | GSK3888130B Dose Level 3 SC | GSK3888130B Dose Level 5 SC
Number analyzed (Participants) | 6 | 6
ng/mL
  DAY 1 (Pre-dose) | NA [NA to NA] — Geometric mean and 95% CI could not be calculated if any values were imputed due to being NQ. | NA [NA to NA] — Geometric mean and 95% CI could not be calculated if any values were imputed due to being NQ.
  DAY 1 (4 Hours) | NA [NA to NA] — Geometric mean and 95% CI could not be calculated if any values were imputed due to being NQ. | 2540.4 [1193.5 to 5407.6]
  DAY 1 (8 Hours) | NA [NA to NA] — Geometric mean and 95% CI could not be calculated if any values were imputed due to being NQ. | 5287.2 [2659.9 to 10509.8]
  DAY 1 (12 Hours) | NA [NA to NA] — Geometric mean and 95% CI could not be calculated if any values were imputed due to being NQ. | 8236.8 [4122.6 to 16456.5]
  DAY 1 (24 Hours) | 1284.2 [795.2 to 2073.7] | 14161.9 [7502.7 to 26731.7]
  DAY 1 (48 Hours) | 2297.0 [1506.7 to 3501.9] | 23239.0 [12191.4 to 44297.5]
  DAY 6 | 3253.7 [2339.4 to 4525.5] | 34612.8 [25180.0 to 47579.2]
  DAY 8 | 3327.1 [2422.0 to 4570.5] | 34801.7 [25828.6 to 46892.0]
  DAY 10 | 3078.4 [2316.4 to 4091.2] | 33654.8 [25702.9 to 44066.9]
  DAY 15 | 2814.4 [2172.0 to 3646.8] | 29870.9 [22782.2 to 39165.2]
  DAY 21 | 2856.1 [2199.3 to 3709.1] | 27433.3 [21634.8 to 34785.7]
  DAY 29 | 2266.1 [1614.4 to 3181.0] | 21108.5 [16241.6 to 27434.0]
  DAY 57 | 1288.8 [817.0 to 2032.9] | 11567.5 [7780.8 to 17197.0]
  DAY 85 | NA [NA to NA] — Geometric mean and 95% CI could not be calculated if any values were imputed due to being NQ. | 5780.9 [3113.3 to 10733.9]

13. Secondary Outcome: Serum Concentrations of GSK3888130B for Dose Levels 6 and 7 IV Administration
Description: as for outcome 11
Time Frame: Day 1: Pre-dose, 30 minutes, 1 hour, 4, 8, 12, 24, 48 hours; Days 6, 8, 10, 15, 21, 29, 57, and 85
Population: Pharmacokinetic (PK) Population. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the 'Overall Number of Participants Analyzed' field. 'Number Analyzed' signifies participants evaluable for the specified time points.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | GSK3888130B Dose Level 6 IV | GSK3888130B Dose Level 7 IV
Number analyzed (Participants) | 9 | 6
ng/mL
  DAY 1 (Pre-dose) | NA [NA to NA] — Geometric mean and 95% CI could not be calculated if any values were imputed due to being NQ. | NA [NA to NA] — Geometric mean and 95% CI could not be calculated if any values were imputed due to being NQ.
  DAY 1 (30 Minutes) | 201271.5 [162241.9 to 249690.2] | 446824.2 [396812.5 to 503139.1]
  DAY 1 (1 Hour) | 365002.7 [300217.9 to 443767.6] | 887258.7 [772728.3 to 1018764.4]
  DAY 1 (4 Hours): number analyzed (Participants) | 8 | 6
  DAY 1 (4 Hours) | 334755.7 [275365.5 to 406955.0] | 845654.2 [743870.4 to 961365.0]
  DAY 1 (8 Hours): number analyzed (Participants) | 8 | 6
  DAY 1 (8 Hours) | 333669.5 [254377.8 to 437677.0] | 839439.2 [725811.5 to 970855.7]
  DAY 1 (12 Hours) | 312692.1 [251461.1 to 388832.9] | 738220.9 [642655.8 to 847997.0]
  DAY 1 (24 Hours) | 288550.5 [235725.2 to 353213.8] | 744312.7 [631579.3 to 877168.5]
  DAY 1 (48 Hours): number analyzed (Participants) | 8 | 6
  DAY 1 (48 Hours) | 221884.4 [173674.6 to 283476.6] | 595269.2 [525651.3 to 674107.3]
  DAY 6 | 186043.0 [154906.8 to 223437.5] | 432475.7 [378277.5 to 494439.2]
  DAY 8 | 148716.7 [122678.0 to 180282.2] | 362540.8 [282254.6 to 465664.2]
  DAY 10 | 150354.6 [119156.0 to 189722.0] | 361427.9 [295704.5 to 441759.0]
  DAY 15 | 124163.7 [104218.9 to 147925.3] | 311912.7 [254633.2 to 382077.2]
  DAY 21 | 108208.1 [95733.2 to 122308.5] | 259786.4 [206492.4 to 326835.0]
  DAY 29: number analyzed (Participants) | 8 | 6
  DAY 29 | 88424.1 [81046.3 to 96473.4] | 207998.2 [147558.4 to 293194.2]
  DAY 57 | 34733.0 [24307.2 to 49630.7] | 100288.2 [65503.1 to 153545.9]
  DAY 85 | 16634.1 [12462.7 to 22201.9] | 53029.2 [34299.5 to 81986.7]

14. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to Time t (AUC[0 to t]) of GSK3888130B for Dose Levels 1, 2 and 4 Intravenous Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3888130B following intravenous administration.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 4, 8, 12, 24, 48 hours; Days 6, 8, 10, 15, 21, 29, 57, and 85
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter(h*ug/mL)
Arm/Group | GSK3888130B Dose Level 1 IV | GSK3888130B Dose Level 2 IV | GSK3888130B Dose Level 4 IV
Number analyzed (Participants) | 3 | 3 | 6
Hours*micrograms per milliliter(h*ug/mL) | 65.81 (75.50) | 1837.01 (48.86) | 13524.34 (16.29)

15. Secondary Outcome: AUC(0 to t) for Dose Levels 3 and 5 Subcutaneous Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3888130B following subcutaneous administration.
Time Frame: Day 1: Pre-dose, 4, 8, 12, 24, 48 hours; Days 6, 8, 10, 15, 21, 29, 57, and 85
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | GSK3888130B Dose Level 3 SC | GSK3888130B Dose Level 5 SC
Number analyzed (Participants) | 6 | 6
h*ug/mL | 3550.71 (38.63) | 35669.70 (25.35)

16. Secondary Outcome: AUC(0 to t) for Dose Levels 6 and 7 Intravenous Administration
Description: as for outcome 14
Time Frame: Day 1: Pre-dose, 30 minutes, 1 hour, 4, 8, 12, 24, 48 hours; Days 6, 8, 10, 15, 21, 29, 57, and 85
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | GSK3888130B Dose Level 6 IV | GSK3888130B Dose Level 7 IV
Number analyzed (Participants) | 9 | 6
h*ug/mL | 153885.4 (12.54) | 387454.3 (24.96)

17. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of GSK3888130B for Dose Levels 1, 2 and 4 Intravenous Administration
Description: as for outcome 14
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 4, 8, 12, 24, 48 hours; Days 6, 8, 10, 15, 21, 29, 57, and 85
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter (ug/mL)
Arm/Group | GSK3888130B Dose Level 1 IV | GSK3888130B Dose Level 2 IV | GSK3888130B Dose Level 4 IV
Number analyzed (Participants) | 3 | 3 | 6
Micrograms per milliliter (ug/mL) | 0.9034 (21.5707) | 4.8156 (18.7069) | 35.6330 (14.4965)

18. Secondary Outcome: Cmax of GSK3888130B for Dose Levels 3 and 5 Subcutaneous Administration
Description: as for outcome 15
Time Frame: Day 1: Pre-dose, 4, 8, 12, 24, 48 hours; Days 6, 8, 10, 15, 21, 29, 57, and 85
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | GSK3888130B Dose Level 3 SC | GSK3888130B Dose Level 5 SC
Number analyzed (Participants) | 6 | 6
ug/mL | 3.4609 (31.2624) | 36.3795 (24.9230)

19. Secondary Outcome: Cmax of GSK3888130B for Dose Levels 6 and 7 Intravenous Administration
Description: as for outcome 14
Time Frame: Day 1: Pre-dose, 30 minutes, 1 hour, 4, 8, 12, 24, 48 hours; Days 6, 8, 10, 15, 21, 29, 57, and 85
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | GSK3888130B Dose Level 6 IV | GSK3888130B Dose Level 7 IV
Number analyzed (Participants) | 9 | 6
ug/mL | 386.4759 (29.7837) | 907.7045 (11.2907)

20. Secondary Outcome: Time to Cmax (Tmax) of GSK3888130B for Dose Levels 1, 2 and 4 Intravenous Administration
Description: as for outcome 14
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 4, 8, 12, 24, 48 hours; Days 6, 8, 10, 15, 21, 29, 57, and 85
Population: as for outcome 12
Measure: Median (Full Range); unit: Hour
Arm/Group | GSK3888130B Dose Level 1 IV | GSK3888130B Dose Level 2 IV | GSK3888130B Dose Level 4 IV
Number analyzed (Participants) | 3 | 3 | 6
Hour | 0.583 [0.55 to 4.00] | 0.550 [0.55 to 4.00] | 0.558 [0.55 to 0.58]

21. Secondary Outcome: Tmax of GSK3888130B for Dose Levels 3 and 5 Subcutaneous Administration
Description: as for outcome 15
Time Frame: Day 1: Pre-dose, 4, 8, 12, 24, 48 hours; Days 6, 8, 10, 15, 21, 29, 57, and 85
Population: as for outcome 12
Measure: Median (Full Range); unit: Hour
Arm/Group | GSK3888130B Dose Level 3 SC | GSK3888130B Dose Level 5 SC
Number analyzed (Participants) | 6 | 6
Hour | 168.000 [120.00 to 222.12] | 143.475 [120.00 to 240.95]

22. Secondary Outcome: Tmax of GSK3888130B for Dose Levels 6 and 7 Intravenous Administration
Description: as for outcome 14
Time Frame: Day 1: Pre-dose, 30 minutes, 1 hour, 4, 8, 12, 24, 48 hours; Days 6, 8, 10, 15, 21, 29, 57, and 85
Population: as for outcome 12
Measure: Median (Full Range); unit: Hour
Arm/Group | GSK3888130B Dose Level 6 IV | GSK3888130B Dose Level 7 IV
Number analyzed (Participants) | 9 | 6
Hour | 1.083 [1.05 to 24.00] | 2.533 [1.05 to 8.00]

23. Secondary Outcome: Half-life (t1/2) of GSK3888130B for Dose Levels 1, 2 and 4 Intravenous Administration
Description: as for outcome 14
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 4, 8, 12, 24, 48 hours; Days 6, 8, 10, 15, 21, 29, 57, and 85
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | GSK3888130B Dose Level 1 IV | GSK3888130B Dose Level 2 IV | GSK3888130B Dose Level 4 IV
Number analyzed (Participants) | 3 | 3 | 6
Hour | 123.73 (35.44) | 633.05 (32.53) | 627.11 (17.66)

24. Secondary Outcome: t1/2 of GSK3888130B for Dose Levels 3 and 5 Subcutaneous Administration
Description: as for outcome 15
Time Frame: Day 1: Pre-dose, 4, 8, 12, 24, 48 hours; Days 6, 8, 10, 15, 21, 29, 57, and 85
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | GSK3888130B Dose Level 3 SC | GSK3888130B Dose Level 5 SC
Number analyzed (Participants) | 6 | 6
Hour | 784.05 (13.62) | 749.02 (31.55)

25. Secondary Outcome: t1/2 of GSK3888130B for Dose Levels 6 and 7 Intravenous Administration
Description: as for outcome 14
Time Frame: Day 1: Pre-dose, 30 minutes, 1 hour, 4, 8, 12, 24, 48 hours; Days 6, 8, 10, 15, 21, 29, 57, and 85
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | GSK3888130B Dose Level 6 IV | GSK3888130B Dose Level 7 IV
Number analyzed (Participants) | 9 | 6
Hour | 563.53 (22.12) | 628.91 (13.71)

26. Secondary Outcome: Clearance (CL) of GSK3888130B for Dose Levels 1, 2 and 4 Intravenous Administration
Description: as for outcome 14
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 4, 8, 12, 24, 48 hours; Days 6, 8, 10, 15, 21, 29, 57, and 85
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliliter per hour (mL/h)
Arm/Group | GSK3888130B Dose Level 1 IV | GSK3888130B Dose Level 2 IV | GSK3888130B Dose Level 4 IV
Number analyzed (Participants) | 3 | 3 | 6
Milliliter per hour (mL/h) | 21.501 (38.138) | 4.240 (52.782) | 6.542 (22.034)

27. Secondary Outcome: Clearance Factor (CL/F) of GSK3888130B for Dose Levels 3 and 5 Subcutaneous Administration
Description: as for outcome 15
Time Frame: Day 1: Pre-dose, 4, 8, 12, 24, 48 hours; Days 6, 8, 10, 15, 21, 29, 57, and 85
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h
Arm/Group | GSK3888130B Dose Level 3 SC | GSK3888130B Dose Level 5 SC
Number analyzed (Participants) | 6 | 6
mL/h | 9.149 (36.810) | 9.297 (27.211)

28. Secondary Outcome: CL of GSK3888130B for Dose Levels 6 and 7 Intravenous Administration
Description: as for outcome 14
Time Frame: Day 1: Pre-dose, 30 minutes, 1 hour, 4, 8, 12, 24, 48 hours; Days 6, 8, 10, 15, 21, 29, 57, and 85
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h
Arm/Group | GSK3888130B Dose Level 6 IV | GSK3888130B Dose Level 7 IV
Number analyzed (Participants) | 9 | 6
mL/h | 5.920 (11.548) | 6.860 (28.592)

29. Secondary Outcome: Number of Participants With Positive Anti-drug Antibodies Against GSK3888130B
Description: Serum samples were collected for the determination of anti-drug antibodies (ADA) using a validated electrochemiluminescent (ECL) immunoassay. The assay involved screening, confirmation and titration steps. If serum samples tested positive in the screening assay, they were considered 'potentially positive' and were further analyzed for specificity using the confirmation assay. Samples that confirmed positive in the confirmation assay were reported as 'positive'. Confirmed positive ADA samples were further characterized in the titration assay to quasi-quantitate the amount of ADA in the sample. Baseline was defined as the latest pre-dose assessment.
Time Frame: Baseline (Day 1), Day 15, Day 29, Day 57 and Day 85
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3888130B Dose Level 1 IV | GSK3888130B Dose Level 2 IV | GSK3888130B Dose Level 3 SC | GSK3888130B Dose Level 4 IV | GSK3888130B Dose Level 5 SC | GSK3888130B Dose Level 6 IV | GSK3888130B Dose Level 7 IV
Number analyzed (Participants) | 15 | 3 | 3 | 6 | 6 | 6 | 9 | 6
Participants
  Baseline (Day 1) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Day 15: number analyzed (Participants) | 15 | 2 | 3 | 6 | 6 | 6 | 9 | 6
  Day 15 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Day 29: number analyzed (Participants) | 15 | 3 | 3 | 6 | 6 | 6 | 8 | 6
  Day 29 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Day 57 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Day 85 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

30. Secondary Outcome: Percent Peak Reduction From Baseline in Derived Free Interleukin 7 (IL 7) in Blood
Description: Free IL-7 levels were derived from total IL-7 and total GSK3888130B concentrations (named as Derived Free IL-7) over time using a nonlinear mixed effects modelling approach. A target-mediated drug disposition model was used to fit the total IL-7 and total GSK3888130B assay concentration data to derive the free-IL-7 concentrations. Peak reduction relative to Baseline (Percent change) was calculated for each participant as; Peak reduction = (1 - minimum [Free IL7/IL7 Baseline])*100. Baseline was defined as the latest pre-dose assessment.
Time Frame: Baseline (Day 1) and up to 8 hours
Population: Pharmacodynamic (PD) Population consisted of all participants in the Safety Population who had at least one post Baseline PD result. Placebo arms were combined as pre-specified in reporting and analysis plan. Zeros reported reflect measured data derived during analysis.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Placebo | GSK3888130B Dose Level 1 IV | GSK3888130B Dose Level 2 IV | GSK3888130B Dose Level 3 SC | GSK3888130B Dose Level 4 IV | GSK3888130B Dose Level 5 SC | GSK3888130B Dose Level 6 IV | GSK3888130B Dose Level 7 IV
Number analyzed (Participants) | 15 | 3 | 3 | 6 | 6 | 6 | 9 | 6
Percent Change | 0.0 (0.00) | 95.8 (1.5383) | 99.1 (0.2841) | 90.3 (4.2311) | 99.9 (0.0246) | 98.6 (0.8138) | 100 (0.0025) | 100 (0.0004)

31. Secondary Outcome: Median Fluorescence Intensity (MdFI) of B-cell Lymphoma 2 (Bcl-2) Expression in CD4+ T Cells in Blood
Description: Blood samples were collected at indicated time points to measure Bcl-2 Expression in CD4+ T Cells as median fluorescence intensity (MdFI). Baseline was defined as the latest pre-dose assessment. MdFI values as a measure of Bcl-2 expression in CD4+ T cells was measured by flow cytometry. Placebo arms were combined as pre-specified in reporting and analysis plan.
Time Frame: Baseline (Day 1) and Day 15
Population: Pharmacodynamic (PD) Population consisted of all participants in the Safety Population who had at least one post Baseline PD result. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in 'Overall Number of Participants Analyzed' field. 'Number Analyzed' signifies participants evaluable for specified time points.
Measure: Median (Full Range); unit: Median fluorescence intensity
Arm/Group | Placebo | GSK3888130B Dose Level 1 IV | GSK3888130B Dose Level 2 IV | GSK3888130B Dose Level 3 SC | GSK3888130B Dose Level 4 IV | GSK3888130B Dose Level 5 SC | GSK3888130B Dose Level 6 IV | GSK3888130B Dose Level 7 IV
Number analyzed (Participants) | 15 | 3 | 3 | 6 | 6 | 6 | 9 | 4
Median fluorescence intensity
  Baseline (Day 1) | 92427.0 [55433 to 114550] | 64576.0 [47010 to 82059] | 68096.0 [54750 to 72379] | 92724.0 [64251 to 104760] | 73182.5 [66900 to 93636] | 93540.5 [79770 to 108965] | 90059.0 [71281 to 118233] | 101786.0 [101255 to 120759]
  Day 15: number analyzed (Participants) | 15 | 2 | 3 | 6 | 6 | 6 | 9 | 4
  Day 15 | 88899.0 [62339 to 128682] | 79882.5 [65395 to 94370] | 75396.0 [53411 to 77550] | 62436.5 [32520 to 77948] | 52592.0 [50096 to 67410] | 55938.5 [26200 to 63447] | 50715.0 [40283 to 65395] | 58098.5 [49364 to 69492]

ADVERSE EVENTS:
Time Frame: All-cause mortality, serious adverse events (SAEs) and common non-serious adverse events (non-SAEs) were collected up to 160 days
Description: All-cause mortality, SAEs and common non-SAEs were reported for the Safety Population which included all participants who received study intervention. Placebo arms were combined as pre-specified in reporting and analysis plan. Dosing information (dosage strengths) has not been disclosed as it is considered as company confidential information (CCI). Dose levels are presented as Dose levels 1 to 7 along with directionality of the dosage within each arm/group.
Arm/Group | Placebo | GSK3888130B Dose Level 1 IV | GSK3888130B Dose Level 2 IV | GSK3888130B Dose Level 3 SC | GSK3888130B Dose Level 4 IV | GSK3888130B Dose Level 5 SC | GSK3888130B Dose Level 6 IV | GSK3888130B Dose Level 7 IV
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/3 | 0/3 | 0/6 | 0/6 | 0/6 | 0/9 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/3 | 0/3 | 0/6 | 0/6 | 0/6 | 0/9 | 0/6
Other Adverse Events (participants affected / at risk) | 8/15 | 3/3 | 2/3 | 6/6 | 2/6 | 4/6 | 8/9 | 5/6
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=15) | GSK3888130B Dose Level 1 IV (N=3) | GSK3888130B Dose Level 2 IV (N=3) | GSK3888130B Dose Level 3 SC (N=6) | GSK3888130B Dose Level 4 IV (N=6) | GSK3888130B Dose Level 5 SC (N=6) | GSK3888130B Dose Level 6 IV (N=9) | GSK3888130B Dose Level 7 IV (N=6)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Swelling face (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected cyst (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood pressure diastolic increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head discomfort (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-03-21): https://cdn.clinicaltrials.gov/large-docs/71/NCT05131971/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-17): https://cdn.clinicaltrials.gov/large-docs/71/NCT05131971/SAP_001.pdf